CLINICAL TRIAL: NCT01676194
Title: Efficacy of Transarterial Chemoembolization With DC-BeadsR Prior to Liver Transplantation for Hepatocellular Carcinoma on Patient Survival : A Prosepctive Multicentre and Randomized Study
Brief Title: Transarterial Chemoembolization Prior to Transplantation for Hepatocellular Carcinoma
Acronym: CATCH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012~A00269-34
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2018-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Transarterial Chemoembolization; Liver transplantation; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-arterial administration of DC BeadsR (Experimental): Intra-arterial administration of DC BeadsR, (1 vial of 100-300 µm) as selectively as possible loaded with doxorubicin (50 mg per procedure) and mixed with an equal volume of contrast medium. The first injection will be performed within 21 days following enlisting and repeated 1-2 times until LT (only if hypervascularized vital tumor tissue is again visible on CT Scan and if liver function remains within Child A stage) or until complete response
  Interventions: Other: Intra-arterial administration of DC BeadsR
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Intra-arterial administration of DC BeadsR
  Arms: Intra-arterial administration of DC BeadsR

SUMMARY:
The hope to treat more patients with hepatocellular carcinoma successfully is however tempered by the shortage of donors leading to an increasing waiting time for liver transplantation (LT). Intention-to-treat analysis have showed that the reported excellent long-term outcome is curtailed and significantly hampered by the growing incidence of patients who must be removed from the waiting list because of tumor progression. A way to face with this issue is to treat hepatocellular carcinoma prior to LT. Among therapeutic options to impede tumor progression, Transarterial Chemoembolization (TACE) is the most common modality used. While there are many studies concerning TACE in this setting, none are controlled studies and thus there is no firm evidence concerning its efficacy in reducing drop-out or increasing survival. Moreover TACE may induce risks (liver failure, arterial complications…) while waiting for LT. Most of the available data have been based upon analysis of patients who received a transplant and have not included patients who were eligible for LT but died, or showed progression, before it could be performed. Therefore, studies conducted on an intention-to-treat basis are needed to clarify the benefit and the risks of TACE prior to LT in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
* Multicentre, prospective, randomized, 2 parallel group study
* Preoperative evaluation of hepatocellular carcinoma in recipients: Tumor diagnosis will be mainly based upon EASL guidelines. HCCs will be classified according to UCSF criteria (size, number of nodules). Clinical and biological status will be updated every 3 month.
* Pre-transplant treatment:

TACE group: An emulsion of Lipiodol and a cytotoxic drug (50mg/m2 of doxorubicin) will be injected as selectively as possible. Then, an embolic agent will be used to assure stop of flow. The first injection will be performed within 10 days following enlisting and repeated every 8 weeks until LT (only if hypervascularized vital tumor tissue is again visible on CT Scan and if liver function remains within Child A stage) or until complete response. Clinical/biological follow-up will be done once a month.

Control group (no treatment until LT): clinical/biological follow-up and CT-scan every 3 month.

This prospective, multicentric, and randomized study may allow investigators to show that TACE with DC-BeadsR can significantly increase intention to treat survival of patients transplanted for HCC. We also expect that this result will be associated with less recurrence of the cancer after transplantation.

Obviously, we expect that the beneficial effect of TACE will be associated with a acceptable rate of complication related to the procedure.

* Pathologic examination: In all patients in whom LT will be performed, the diagnosis of hepatocellular carcinoma will be confirmed by a histological examination of the explanted liver.
* Dropout criteria: Patients with progression but still meeting the transplant criteria will be maintained in their respective group. Patients with progression over the transplant criteria will be excluded from the waiting list and censored.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years
* With well compensated cirrhosis and hepatocellular carcinoma meeting UCSF criteria
* Without general contraindication to LT
* Written informed consent.

Exclusion Criteria:

* Patients that already had TACE
* Or other local treatment for HCC
* Or neoadjuvant systemic chemotherapy
* Or planned living donor
* Or non arterialized lesion(s)
* Or Contraindication to DC-BeadsR
* Or allergy to contrast agents
* Or contraindication to Doxorubicin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05-28 (Actual); Study Completion 2016-02-16 (Actual)

PRIMARY OUTCOMES:
Survival | 3 years
  Intention to treat survival at 3 years following inscription on the waiting list for liver transplantation in patient with hepatocellular carcinoma

SECONDARY OUTCOMES:
Dropout rate | 3 years
  Dropout rate (tumor progression beyond transplanted criteria and all causes mortality)
Post-transplantation survival rate | 3 years
Allograft survival | 3 years
Time to dropout | 3 years
Recurrence rate | 3 years
TACE-induced complications (local and general) | 3 years
Contrast agent - induced complications | 3 years
Doxorubicin-induced complications | 3 years
Efficacy of TACE | 3 years
  Efficacy of TACE (morphological response to TACE: captation rate of Lipiodol and morphological response (RECIST guidelines), as well as histological criteria: percentage of necrosis on pathological examination)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe COMPAGNON, MD, Principal Investigator — Service de Chirurgie Digestive - Transplantation Hépatique / Hôpital Henri Mondor - Assistance Publique-Hôpitaux de Paris / Faculté de Médecine - Université Paris-Est; Karim BOUDJEMA, MD PhD, Principal Investigator — Service de Chirurgie Hépato-biliaire et Digestive, Transplantation Hépatique / CHU de Rennes / Université de Rennes 1; Bruno Laviolle, MD, PhD, Study Chair — Service de Pharmacologie et CIC - INSERM 0203 / CHU de Rennes / Université de Rennes
Locations (7):
- France (7):
  - Hôpital Henri Mondor - Assistance Publique-Hôpitaux de Paris, Créteil
  - Hôpital Michalon, CHU de Grenoble, Grenoble
  - Hôpital Claude Huriez, CHU de Lille, Lille
  - Hôpital de la Croix Rousse, HCL, Lyon, Lyon
  - Hôpital Saint-Antoine / APHP, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Trousseau, CHU de Tours, Tours